CLINICAL TRIAL: NCT00672113
Title: Effects of Adalat LA 30 mg and Coracten 30 mg on Nifedipine Plasma Concentration , Plasma Catecholamines, Blood Pressure Response and Heart Rate in Fed Mild to Moderate Hypertensive Patients.
Brief Title: Effects of Adalat LA and Coracten on Drug Levels, Blood Pressure, and Heart Rate in Fed Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 100128
Record Dates: First submitted 2008-04-16; First posted 2008-05-06 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Adalat (Nifedipine, BAYA1040)
- Arm 2 (Active Comparator)
  Interventions: Drug: Coracten

INTERVENTIONS:
Drug: Adalat (Nifedipine, BAYA1040) — Nifedipine GITS 30 mg followed by Coracten 30 mg then back to nifedipine GITS 30 mg
  Arms: Arm 1
Drug: Coracten — Coracten 30 mg followed by nifedipine GITS 30 mg then back to Coracten 30 mg
  Arms: Arm 2

SUMMARY:
This study compares the effect of Adalat LA to Coracten on drug levels as well as changes in blood pressure and heart rate in fed hypertensive subjects. Subjects are dosed with either Adalat or Coracten for first 2 weeks, followed by the other drug for 2 weeks, and then switched back to the original drug for one day. Blood samples, blood pressure, and heart rate are taken before and after each treatment period.

ELIGIBILITY:
Inclusion Criteria:- Mild to moderate hypertension (sitting DBP > 95 - <114 mmHg and/or SBP > 140 - < 160 mmHg) currently untreated. or- Previously diagnosed mild to moderate hypertension (DBP 95-114 mmHg and/or SBP 140 - 160 mmHg) well controlled on current treatment but experiencing adverse events who can be safely switched to the study treatments. or- Previously diagnosed mild to moderate hypertension (DBP 95-114 mmHg and/or SBP 140 - 160 mmHg), well controlled on current treatment, without adverse events, and willing to participate in the study. Exclusion Criteria:- Females who are pregnant, nursing or of childbearing age, unless sterilised. Subjects receiving any form of contraception are not eligible.- Subjects with a medical history of cardiac disease within 6 months (e.g. myocarditis or pericarditis, aortic stenosis, myocardial infarction, unstable angina pectoris or severe angina pectoris). - Subjects with history or evidence of congestive heart failure- Subjects with evidence of clinically important arrhythmia or conduction disturbances requiring treatment.- Subjects with severe liver disease (liver enzymes twice the upper limit of "normal") or other gastrointestinal (GI) tract diseases including inflammatory bowel disease or Crohns disease- Subjects with lactose intolerance.- Subjects with renal diseases (creatinine > 1.5 mg/dL), which could alter the absorption, metabolism or excretion of the study drugs.- Subjects with Type I diabetes. - Subjects taking drugs which may interfere with the metabolism of nifedipine (cimetidine, ranitidine, quinidine, digoxin, rifampicin, diltiazem, cisapride, quinupristin/dalfopristin, cyclosporin, phenytoin or other antiepileptic drugs,).- Subjects suffering from secondary or malignant hypertension.- Subjects with any known contraindication (e.g. hypersensitivity) to nifedipine or other calcium channel blockers of the dihydropyridine class.- Subjects with previously known clinically significant abnormalities of laboratory tests that might suggest further investigation.- Subjects with a resting heart rate < 50 bpm or > 100 bpm.- Subjects with a history of drug and/or alcohol abuse.- Subjects unwilling to comply with the protocol.- Subjects who have participated in another clinical trial within the last month.- Subjects with neurologic or psychiatric illness requiring medication (e.g. tricyclic antidepressants, MAO inhibitors).- Subjects with clinical evidence of ongoing or recent (within the last year) stroke or transient ischemic attacks.- Subjects with pre-existing severe gastrointestinal or oesophageal constriction or narrowing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-12; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Maximum change in plasma norepinephrine in fed state dose administration to within 6 hours after the first dose | Up to 6 hours after first dose

SECONDARY OUTCOMES:
Single dose: change in epinephrine, SBP, DBP, HR, and plasma nifedipine concentration time profile including Cmax and tmax under fed conditions | After first dose
Multi-dose: the change in norepinephrine, epinephrine, SBP, DBP, HR, and plasma nifedipine concentration time profile including Cmax and tmax under fed conditions | After 2 weeks dosing
The switch: the change in norepinephrine, epinephrine, SBP, DBP, HR, and plasma nifedipine concentration time profile including Cmax and tmax under fed conditions after switching from Coracten to nifedipine and vice versa | Week 2 plus 1 day to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cambridge, Cambridgeshire, United Kingdom